CLINICAL TRIAL: NCT06353815
Title: Clinical Evaluation of Anaesthetic Efficacy of 4% Articaine Buccal Infiltration Versus Inferior Alveolar Nerve Block for Restorative Dental Treatment in Mandibular First Permanent Molars: A Randomized Clinical Tria
Brief Title: Clinical Evaluation of Anaesthetic Efficacy of 4% Articaine Buccal Infiltration Versus Inferior Alveolar Nerve Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Moustafa, Resident at Pediatric Dentistry Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: anaesthetic efficacy
Record Dates: First submitted 2024-03-31; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Restorative Dental Treatment by Buccal Infiltration Anaesthesia
Keywords: buccal infiltration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental group) 4% articaine infiltration (Experimental)
  Interventions: Other: 4% articaine infiltration
- Group II (Control group) 4% articaine inferior alveolar nerve block (Active Comparator)
  Interventions: Other: 4% articaine infiltration

INTERVENTIONS:
Other: 4% articaine infiltration — Two injections using short needle and dental syringe will be given , the first injection is 1.5 ml out of 1.8 ml of 4% articaine with 1:100,000 epinephrine (ARTINIBSA 4% 1:100,000) in the mucobuccal fold adjacent to the mandibular first Molar, the second injection is 0.3 ml in the lingual side for lingual soft and hard tissues .

SUMMARY:
Clinical evaluation of anaesthetic efficacy of 4% articaine buccal infiltration versus inferior alveolar nerve block during restorative dental treatment in mandibular first permanent molars

ELIGIBILITY:
Inclusion Criteria:

* Clinical Criteria:

  * Children aged between 6 years and 9 years having:
  * Mandibular first permanent molar with simple caries not involving pulp showing the following criteria: A. No history of spontaneous pain, pathologic mobility, draining sinus tract, redness or swelling of the vestibule. B. Normal gingival and periodontal condition, with no sensitivity to vestibular palpation, and no pain on percussion test.

Radiographic criteria:

* No sign of radiolucency in periapical or furcation area.
* No widening of PDL space or loss of lamina dura continuity.
* No evidence of internal/external pathologic root resorption

Exclusion Criteria:

* • Uncooperative children.

  * Children with systemic disease.
  * Lack of informed consent by the child patient's parent.
  * Refusal of participation.
  * Allergy from anesthetic agent.
  * Acute infection

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Success of local anesthesia | 10 minutes
  Operator will record the LA as Successful if the scheduled restorative treatment was completed with standard treatment management strategies after administration of the trial anaesthetic. If treatment could not be continued after 10 minutes from when the LA was first administered, and the full 1.8 ml cartridge of the trial anaesthetic had been used, then the LA was considered unsuccessful

SECONDARY OUTCOMES:
Child behavior during treatment | Intraoperative
  Doaa Moustafa: he patient's behavior will be evaluated for pain perception during treatment using the SEM scale (Appendix 3: SEM scale ). The SEM scale is an objective pain [10:04 pm, 31/3/2024] Doaa Moustafa: assessment scale with scores ranging from 1 to 4, illustrating comfort to severe discomfort based on sounds, eye, motor parameters

IPD SHARING:
Plan to Share IPD: Undecided